CLINICAL TRIAL: NCT02309723
Title: A Survey of Clinicians to Assess the Influence of Beta-amyloid Imagining Information on the Diagnosis and Management of Hypothetical Patients With Cognitive Complaints
Brief Title: Influence of Beta Amyloid Imaging on Care of Patients Cognitive Complaints.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CEVR-2013-001
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Neuroimaging; Diagnostic Tool
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

ARMS (3):
- Positive beta amyloid findings (Experimental): Beta amyloid imaging results indicated a positive finding.
  Interventions: Device: Beta amyloid imaging
- Negative beta amyloid findings (Experimental): Beta amyloid imaging results indicated a negative finding.
  Interventions: Device: Beta amyloid imaging
- No beta amyloid information (No Intervention)

INTERVENTIONS:
Device: Beta amyloid imaging
  Arms: Negative beta amyloid findings; Positive beta amyloid findings

SUMMARY:
When older patients develop cognitive problems - like memory loss - there may be any of several underlying causes, sometimes occurring in combination. Clinicians have a better chance of providing appropriate treatment if they understand what the cause of the problem is. A diagnostic tool can help the patient by helping the clinician to make a more accurate diagnosis. This study investigates whether a new diagnostic tool - beta amyloid imaging - may potentially improve medical practice. The tool can potentially improve practice only if it can influence clinical judgment. This study investigates whether the provision of beta amyloid imaging information influences clinical judgment. The investigators will conduct a survey that presents clinicians with descriptions of hypothetical older patients with cognitive complaints. Some of the respondents also receive beta amyloid imaging information. The investigators will test the investigators hypothesis that the information will affect diagnostic judgment and management recommendations by comparing the responses of clinicians who receive the beta amyloid information to the responses of clinicians who do not.

ELIGIBILITY:
Inclusion Criteria:

* Practicing clinicians describing their training and practice as any of the following: neurologist, geriatrician, psychiatrist.
* Included respondents must also attest that they are a physician who is experienced in the assessment and diagnosis of dementia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T. Cohen, Ph.D, Study Director — Tufts Medical Center; Peter J Neumann, ScD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Beta Amyloid Findings: Beta amyloid imaging results indicated a positive finding.
  Beta amyloid imaging
- Negative Beta Amyloid Findings: Beta amyloid imaging results indicated a negative finding.
  Beta amyloid imaging
Period: Overall Study
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information
Started | 129 | 128 | 129
Completed | 105 | 105 | 105
Not Completed | 24 | 23 | 24
Not completed — Withdrawal by Subject | 24 | 23 | 24

BASELINE CHARACTERISTICS:
Population: number of clinicians responded to the email
Groups:
- Positive Beta Amyloid Findings: Survey respondents presented scenario in which beta amyloid imaging results indicated a positive finding.
- Negative Beta Amyloid Findings: Survey respondents presented scenario in which beta amyloid imaging results indicated a negative finding.
- No Beta Amyloid Information: Survey respondents presented scenario with no beta amyloid information.
- Total: Total of all reporting groups
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information | Total
Number analyzed (Participants) | 106 | 105 | 104 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are reported by subject.
  years | 51.3 (8.8) | 51.5 (7.8) | 52.7 (8.0) | 51.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 87 | 134
  Male | 82 | 82 | 17 | 181
Beta Amyloid imaging findings [Number; unit: participants] | 106 | 105 | 104 | 315

OUTCOME MEASURES:

1. Primary Outcome: Influence of the Neuroimaging Test on a Finding of Alzheimer's Disease as the Underlying Cause of the Mild Memory Loss
Description: Proportion of respondents who identify Alzheimer's Disease as the sole or a contributing factor that is responsible for the patient's cognitive complaint.
Time Frame: Online Survey - completion during the estimated 2-3 month field period
Measure: Number; unit: participants
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information
Number analyzed (Participants) | 105 | 106 | 104
participants
  Diagnosis confidence: not at all confident | 3 | 12 | 9
  Diagnosis confidence: somewhat confident | 31 | 34 | 30
  Diagnosis confidence: confident | 43 | 38 | 46
  Diagnosis confidence: very confident | 25 | 18 | 14
  Diagnosis confidence: extremely confident | 3 | 4 | 5

2. Primary Outcome: Likelihood of Recommending a Medication Indicated for Alzheimer's Disease
Description: Proportion of respondents who recommend a medication indicated for the treatment of Alzheimer's Disease, including Acetylcholinesterase inhibitors, N-methyl-D-aspartate receptor antagonists, Typical antipsychotics - e.g., Chlorpromazine (Thorazine), Haloperidol (Haldol), Atypical antipsychotics - e.g., Clozapine (Clozaril), Risperidone (Risperdal), Antidepressant - e.g., Citalopram (Celexa), Venlafaxine (Effexor), Antianxiety agent - e.g. Benzodiazepines, Buspirone (Buspar).
Time Frame: Online Survey - completion during the estimated 2-3 month field period
Measure: Number; unit: participants
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information
Number analyzed (Participants) | 106 | 105 | 104
participants | 93 | 76 | 92

3. Primary Outcome: Likelihood of Recommending That Spouse Take Various Cognitive Deficit Disease Management Measures
Description: Proportion of respondents who recommend that the patient's spouse take actions that would be appropriate if the patient has Alzheimer's disease, including: (1) discussion of advance care planning, (2) monitoring of patient's finances, (3) assessment of how compatible the patient's job is with his conditions, (4) the initiation of precautions to ensure the patient is properly taking his medications to manage hypertension and hyperlipidemia.
Time Frame: Online Survey - completion during the estimated 2-3 month field period
Measure: Number; unit: participants
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information
Number analyzed (Participants) | 106 | 105 | 104
participants | 67 | 61 | 66

ADVERSE EVENTS:
Arm/Group | Positive Beta Amyloid Findings | Negative Beta Amyloid Findings | No Beta Amyloid Information
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/105 | 0/104
Other Adverse Events (participants affected / at risk) | 0/106 | 0/105 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No